CLINICAL TRIAL: NCT06840444
Title: The Firefly Mobile App: A Digital Health Solution for Healthy Sleep in Teens
Brief Title: Implementation & Dissemination of a Digital Health Intervention for Adolescent Sleep
Acronym: Firefly
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00161292
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Insomnia; Adolescent; Digital Health
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Teen Advisory Board (TAB)/Beta Cohort 1: These teens will co-design and beta-test an app prototype.
  Interventions: Behavioral: Firefly Mobile App: A Digital Health Solution for Healthy Sleep in Teens
- Beta Cohort 2: These teens will do the second round of beta-testing for the app prototype.
  Interventions: Behavioral: Firefly Mobile App: A Digital Health Solution for Healthy Sleep in Teens

INTERVENTIONS:
Behavioral: Firefly Mobile App: A Digital Health Solution for Healthy Sleep in Teens — A six week cognitive behavioral therapy for insomnia program delivered via a mobile app.

SUMMARY:
The goal of this study is to form a Teen Advisory Board (TAB), who will partner with our study team to co-design a beta-test a new prototype of the Firefly program, a mobile-native insomnia cognitive behavioral therapy intervention for teens. This new prototype will have addressed issues that adolescents who had used the first version of the program deemed to be barriers to engaging with the treatment.

DETAILED DESCRIPTION:
The aims of this study are to: 1) form a Teen Advisory Board (TAB) of teens with self-reported insomnia symptoms, 2) co-design a functional app prototype for sleep with TAB, 3) conduct two rounds of beta-testing to inform the iterative refinement of the app prototype. Participants will include 40 youth and their parents; 10 youth will participate in the TAB and first round 1 of beta-testing, and a separate cohort of 30 youth will participate in a second round of beta-testing. Youth will be ages 13-18 years and will have self-reported insomnia symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 13-18 years old
* Self-reported insomnia symptoms

Exclusion Criteria:

* Non-English speaking

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Youth with self-reported insomnia symptoms, aged 13-18.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Program Completion Percentage | Immediately post-treatment

SECONDARY OUTCOMES:
Treatment Acceptability Ratings | Immediately post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Kansas University Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes